CLINICAL TRIAL: NCT01461746
Title: A Phase II Trial of Docetaxel/Cisplatin Chemotherapy Followed by Pelvic Radiation Therapy in Patients, With High-risk Endometrial Carcinoma After Staging Surgery
Brief Title: Efficacy Study of Chemotherapy Followed by Radiation Therapy to Treat Endometrial Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Joo-Hyun Nam, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANSGOG-001
Record Dates: First submitted 2011-10-24; First posted 2011-10-28 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Docetaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherpay and radiation therapy (Experimental): Docetaxel plus cisplatin followed by radiation therapy
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 70mg/m2BSA, q 3 weeks, 3 cycles
Drug: Cisplatin — Cisplatin 60mg/m2BSA, q 3 weeks, 3 cycles
Radiation: Radiation therapy — Pelvic radiation therapy (Extended filed radiation therapy and addition of brachytherapy is allowed)

SUMMARY:
Previous some studies suggested the addition of chemotherapy to radiation therapy after surgery may have survival benefit in patients with high risk endometrial cancer. In addition, docetaxel plus cisplatin regimen may have similar efficacy with paclitaxel plus carboplatin which is currently used in most cases. However, docetaxel plus cisplatin may cause less toxicity compared to paclitaxel plus carboplatin. Therefore, the investigators aimed to analyze the efficacy of docetaxel plus cisplatin regimen followed by radiation therapy after surgery in patients with high risk endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* One of following high risk groups Stage III after staging operation Stage II (Type I hysterectomy + BSO + LND) Stage I + two of [Grade III, LVSI+, Mm>1/2] Clear cell or serous carcinoma: stage IB-II
* Age: 20-75
* ECOG PS: 0-2
* Adequate organ function BM: WBC ≥ 3,000/mm3, ANC≥1,500/mm3, Plt≥100X103/mm3, Hb≥10.0 g/dl Kidney: Creatinine <1.25 × UNL이고, GFR ≥ 60 Liver: AST, ALT< 3×UNL, T- bil<1.5 mg/ mm3
* Informed Consent

Exclusion Criteria:

* Previous chemotherapy or pelvic RT
* Hormone therapy within 4 weeks
* Other malignant disease
* Uncontrolled medical disease
* Infection requiring antibiotics
* Symptomatic CHF, RF, Angina, Arrhythmia, etc.
* Neurosis or psychosis
* Etc.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2011-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years after completion of study treatment

SECONDARY OUTCOMES:
Overall survival | 2 years after completion of study treatment
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Before each chemotherapy, an expected average of 3 weeks
Quality of life | 3 months after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hyun Nam, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea